CLINICAL TRIAL: NCT05609331
Title: Feasibility, Safety, and Efficacy of Stereotactic MRI-Guided Adaptive Radiation Therapy (SMART) for Central Lung Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: <75 % participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0371; NCI-2022-09313 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-10-28; First posted 2022-11-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage I-(Simulated Online Adaptive Planning) (Experimental): Participants will receive treatment with the conventional CT-based radiation therapy and receive additional MRI scans.
  Interventions: Other: Simulated Online Adaptive Planning
- Stage II (Stereotactic MRI-guided adaptive radiotherapy-SMART) (Experimental): Participants will receive treatment with the investigational MRI-guided radiation therapy.
  Interventions: Radiation: Stereotactic MRI-guided adaptive radiotherapy-SMART

INTERVENTIONS:
Other: Simulated Online Adaptive Planning — The results of the MRI-guided radiation therapy will be compared to conventional radiation therapy (guided by CT scans) during this study
  Arms: Stage I-(Simulated Online Adaptive Planning)
Radiation: Stereotactic MRI-guided adaptive radiotherapy-SMART — The results of the MRI-guided radiation therapy will be compared to conventional radiation therapy (guided by CT scans) during this study
  Arms: Stage II (Stereotactic MRI-guided adaptive radiotherapy-SMART)

SUMMARY:
To learn if using MRI (magnetic resonance imaging) to guide radiation therapy can help to control central lung cancer. The results of the MRI-guided radiation therapy will be compared to conventional radiation therapy (guided by CT scans) during this study.

DETAILED DESCRIPTION:
Primary Objective:

Stage I: Assess the feasibility of SMART for central lung tumors with simulated online adaptive planning.

Stage II: Evaluate the feasibility and safety of SMART in central lung tumors treated with 50Gy in 4-5 fractions.

Secondary Objectives:

Stage I: Determine clinical features that predict for greater benefit from adaptive planning Stage I: Determine the potential dosimetric benefit of SMART for central lung tumor Stage II: Determine the safety and efficacy of SMART for central lung tumors treated with 50Gy in 4-5 fractions.

Exploratory objectives:

Validate cine imaging and motion management strategies on the MR-linac

ELIGIBILITY:
Stage I:

Inclusion Criteria:

1. Primary lung cancer or lung metastasis from another primary
2. Central tumors ≤ 2 cm from any mediastinal critical structure (proximal bronchial tree, esophagus, heart, brachial plexus, major vessels, spinal cord, phrenic nerve, and recurrent laryngeal nerve
3. Age ≥ 18 years
4. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

1. Contraindications to MR imaging (e.g. implanted metallic prostheses, defibrillators, stimulators, pacemakers, or neurotransmitters) per institutional policy on management of patients with internal and external medical devices
2. Inability to tolerate MR imaging (Ie. history of claustrophobia)
3. Women who are pregnant. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.

Stage 2:

Inclusion Criteria:

1. Primary lung cancer or lung metastasis from another primary
2. Central tumors ≤ 2 cm from any mediastinal critical structure (proximal bronchial tree, esophagus, heart, brachial plexus, major vessels, spinal cord, phrenic nerve, and recurrent laryngeal nerve
3. Age ≥ 18 years
4. Ability to understand and the willingness to sign a written informed consent
5. Determined by two thoracic radiation oncologists to require > 10-15 fraction regimens if treated with CT-based, non-adaptive radiation therapy

Exclusion Criteria:

1. Contraindications to MR imaging (e.g. implanted metallic prostheses, defibrillators, stimulators, pacemakers, or neurotransmitters) per institutional policy on management of patients with internal and external medical devices
2. Inability to tolerate MR imaging (Ie. history of claustrophobia)
3. Women who are pregnant. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0, Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Saumil Gandhi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M. D. Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT05609331/ICF_001.pdf